CLINICAL TRIAL: NCT05546983
Title: How to Report Postoperative Outcomes After a Paediatric Cardiac Surgery ?
Acronym: Pedia-Card
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8717
Record Dates: First submitted 2022-09-15; First posted 2022-09-21 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Congenital Heart Disease in Children
Keywords: Congenital Heart Disease; Abnormality in newborns
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Congenital heart disease is a common abnormality in newborns. The marked improvement in the surgical management of congenital heart disease has led to a reduction in postoperative mortality, historically a quality criterion for surgical and resuscitation management. With the improvement of medical knowledge and surgical techniques, mortality is no longer a single quality criterion for a center and the search for other quality criteria is essential.

ELIGIBILITY:
Inclusion criteria:

* Minor patients, under the age of 18
* operated at the HUS between 01/01/2010 and 03/31/2022 for transposition surgery of the great vessels (arterial switch) with or without CIV; or isolated ventricular septal closure
* Child or holders of parental authority who do not object to the reuse of their data for scientific research purposes.

Exclusion criteria:

* Transposition surgery of the great vessels associated with coarctation of the aorta, pulmonary stenosis or any other complex malformation
* Surgical technique different from the arterial switch for the transpositions of the great vessels
* Closure of interventricular communication associated with another complex heart malformation (tetralogy of Fallot, atrioventricular canal, right ventricle with double outlet, etc.)
* Child or holders of parental authority who have expressed their opposition to the reuse of their data for scientific research purposes.

Ages: 1 Year to 17 Years | Sex: All
Age Groups: Child
Study Population: Minor patients, under the age of 18 operated at the HUS between 01/01/2010 and 03/31/2022 for transposition surgery of the great vessels (arterial switch) with or without CIV; or isolated ventricular septal closure
Sampling Method: Non-Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Retrospective analysis of the quality criteria described in the literature after pediatric cardiac surgery by studying their behavior within a local cohort within the University Hospitals of Strasbourg | Files analysed retrospectively from January 01, 2010 to March 31, 2022 will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Pédiatrie 1 - CHU de Strasbourg - France, Strasbourg, France